CLINICAL TRIAL: NCT03728595
Title: A Predictive Score to Reduce the Use of Hypoxic-altitude Simulation Test (HAST) in Patients With Chronic Respiratory Disease Planning Air Travel - an External Validation Prospective Study
Brief Title: Validation of a Predictive Score for HAST
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RM18/109075; 247902 (Other: IRAS); 18/WS/0117 (Other: HRA/REC4 West of Scotland)
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Chronic Respiratory Disease; Hypoxia, Altitude; COPD; ILD; Cystic Fibrosis
Keywords: gas exchange; in-flight hypoxia; hypoxic altitude simulation test; blood gas response
MeSH Terms: conditions — Altitude Sickness; Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis | interventions — Blood Specimen Collection; Spirometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The Investigator will collect a blood sample to be processed for serum bicarbonate.
  As processing a sample for serum bicarbonate is very susceptible to pre-analytical sources of error, samples will be analysed immediately after collection and then discarded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lung disease having HAST: Patients with chronic respiratory diseases who had a hypoxic altitude simulation test (HAST) for clinical purposes will have for research purposes:
  * venepuncture
  * spirometry.
  Interventions: Diagnostic Test: Venepuncture; Diagnostic Test: Spirometry; Diagnostic Test: Hypoxic altitude simulation test (HAST)

INTERVENTIONS:
Diagnostic Test: Venepuncture — A blood sample will be taken for serum bicarbonate
Diagnostic Test: Spirometry — All patients who have not had a spirometry in the 12 months prior to the HAST will undergo one on the day of the HAST.
Diagnostic Test: Hypoxic altitude simulation test (HAST) — HAST will be performed as per clinical team request. No changes to this intervention will be made for research purposes.

SUMMARY:
Patients with chronic lung diseases travelling by plane often suffer with symptoms related to lower oxygen levels they are exposed to while flying.

Therefore, patients with respiratory conditions are routinely assessed to establish if they need supplemental oxygen in flight. A hypoxic altitude simulation test (HAST) is often part of this assessment and consists in having patients breathe a oxygen/nitrogen blend with a lower oxygen concentration compared to normal room air, simulating in-flight conditions. Oxygen levels are measured before and after the test through a blood sample (from the earlobe or an artery in the wrist) and with a finger probe. In-flight oxygen is required if the oxygen level in the blood is lower than 6.6 kPa. HASTs are time consuming, costly, and require a dedicated hospital appointment.

Using historical data, the Investigators developed scores based on capillary blood gas (blood sample from the earlobe), diagnosis and sex to predict the outcome of the HASTs. The Investigators validated the proposed scores in a separate historic cohort of patients and showed it had good concordance with the HASTs results.

In this study, the Investigators want to confirm prospectively if the score, based on blood results (venous and/or earlobe), can predict the outcome of the HASTs and therefore reduce the number of tests performed, travel time for patients, and costs for the NHS.

All patients, aged 18 or older, who are having a HAST for clinical purposes at the cardio-respiratory lab at Leeds Teaching Hospital NHS Trust will be invited to take part in the study. The Investigators will record diagnosis, results of HAST and previous spirometry from the medical notes, perform a spirometry if not done in the previous 12 months and collect a blood sample (one tube, 4 mls). With these data, the Investigators will calculate the score and assess its agreement with the outcome of the HAST.

Each participant's involvement in the study will last for approximately 90-120 minutes, which is the normal duration of a HAST.

The Investigators aim to include up to 280 subjects in the study.

DETAILED DESCRIPTION:
Over the last two decades, there has been a significant increase in the number of people flying on a regular basis. As a result, more individuals with chronic respiratory disease are being referred for formal assessment to assess if they require inflight oxygen.

At cruising altitude, passengers are exposed to reduced atmospheric pressure equivalent to an altitude of 8000 ft, corresponding to a reduction of oxygen from 21% to approximately 15%. National and International recommendations on air travel suggest screening patients with chronic lung diseases for the need of in-flight oxygen supplementation. However, due to the paucity of available evidence, there is no consensus on which investigation should be performed and the precise risk factors associated with in-flight complications.

The British Thoracic Society, which published the most recent and comprehensive recommendations on this topic, recommends that patients with respiratory diseases should be assessed clinically, and in specific situations, a hypoxic altitude simulation tests (HAST) should be performed. Unfortunately, the vast majority of these recommendations are level C at best, as current evidence is limited to a handful of prospective or retrospective analyses.

A standard hypoxic altitude simulation test requires the patients to breathe a blend of 15% oxygen in nitrogen for 20 minutes. This simulates the oxygen tension at 8000 ft, the equivalent cabin pressure. Blood gas measurements are taken before and after the test. A fall in the pO2 below 6.6 kPa is considered indicative for use of in-flight oxygen.

Often the HASTs yield negative results (i.e. no inflight oxygen required). These tests are heavy on resources, time consuming, costly, not widely available and require dedicate hospital appointment. Thus, predictors of outcomes of HASTs are needed to reduce the number of HASTs performed.

Several studies have looked at predictors of oxygen desaturation during HAST in varying populations with the aim of better selecting patients who need the test. However, results have been inconclusive. Data on the role of baseline oxygenation, FEV1 and exercise test in predicting oxygen desaturation during the HAST are conflicting and most studies have been too small to provide decisive answers.

The Investigators recently developed and validate, on historical data, three scores to predict negative HASTs, according to the BTS 2011 recommendations (i.e. scores predicting which patients do not need to undergo a formal assessment). All of these had good ROC AUC and agreement with the outcome of the HAST in the retrospective dataset.

The Investigators hypothesise that the multivariable score (Model 1), based on a combination of CBG variables (bicarbonate and oxygen saturation) and baseline diagnosis (ILD and COPD) would be the best predictor of negative response in a formal HAST. Furthermore, the Investigator hypothesise that the score could be further simplified for the use in clinical practice by measuring the serum bicarbonate and oxygen saturation through a pulse oximeter (Model 1s). This is in light of the good arterio-venous concordance previously demonstrated for bicarbonate and of the good reliability of non-invasive measurement of oxygen saturation. Such a simplified score, if its predictive value is confirmed, would not only reduce the number of unnecessary HAST performed, but also minimise patients' discomfort and hospital appointments, reducing the costs for the NHS.

In this prospective single centre study, the Investigators will assess the validity of the best performing score (Model 1) derived in our retrospective study for negative HAST. In addition, the Investigators want to verify whether the use of SpO2 in place of SO2 and of serum bicarbonate in place of capHCO3 would allow for similar results. The investigators also aim to evaluate the performance of the other predictive scores previously derived in our retrospective analysis, and, if none of these models are a good and effective predictor, we aim to develop a new model based on newly measured data.

The Investigators aim to enroll up to 280 subjects, but interim analyses will be performed with the scope to early terminate the study if primary outcome is met.

Demographic and baseline characteristics of patients will be analysed on the whole population and by the cohorts depending on the underlying diagnosis and the outcome of the HAST.

Receiver operating characteristics (ROC) curves will be plotted to test the hypothesis that the scores are good predictors of negative HASTs. Diagnostic values of the scores will be expressed by sensitivity, specificity, positive and negative predictive values.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old (at the time of HAST)
* Clinically stable
* Hypoxic altitude simulation test, scheduled as part of the clinical care

Exclusion Criteria:

* Inability to provide informed consent
* Being part of a clinical trial, which would exclude patients who are taking part in other studies including observational studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient attending for a HAST at Leeds Teaching Hospital NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
ROC AUC for Model 1 (3*SaO2 - HCO3 - 4 if ILD - 4 if F -3 if COPD), and the relative sensitivity, specificity, positive and negative predictive value of the threshold identified for negative and positive HAST | Up to 36 months
  The score based on Model 1 will be computed for all subjects and ROC curve analyses will be used to assess predictive value. Sensitivity, specificity, PPV and NPV for criteria previously identified in a historic cohort will be assessed.

SECONDARY OUTCOMES:
ROC AUC for the simplified score (3*SpO2 - sHCO3 - 4 if ILD - 4 if F - 3 if COPD) | Up to 36 months
  The simplified score will be computed for all subjects. ROC analyses will be performed and criteria to identify negative and positive HAST at 95%, 97.5% and 99% will be chosen.
ROC AUC for Model 2, and Model 3 and for baseline pO2 and relative sensitivity, specificity, positive and negative predictive value of the previously identified thresholds. | Up to 36 months
  The scores based on Model 2 and 3 will be computed for all subjects and ROC curve analyses will be used to assess predictive value. Sensitivity, specificity, PPV and NPV for criteria previously identified in a historic cohort will be assessed.

OTHER OUTCOMES:
Negative and positive predictive value for the criteria chosen for the simplified score. | Up to 36 months
  Criteria to maximise specificity for negative and positive HAST, respectively, will be chosen for the simplified score (Outcome 2). NPV and PPV for these criteria will be assessed.
Identification of a new predictive model for the outcome of the HAST | Up to 36 months
  Exploratory outcome: in case the previously identified models will not be validated, a new score will be developed using binary logistic regression analysis.
Identification of a model to predict the flow-rate of oxygen required by patients who have a positive HAST. | Up to 36 months
  During the HAST flow-rate of oxygen is titrated for patients with a positive outcome. As exploratory outcome we aim to develop a model to predict the final flow-rate required for patients who need oxygen in flight.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Spoletini, Principal Investigator — Leeds Teaching Hospital NHS Trust
Locations (1):
- St James's University Hospital, LTHT, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aerospace Medical Association; Aviation Safety Committee; Civil Aviation Subcommittee. Cabin cruising altitudes for regular transport aircraft. Aviat Space Environ Med. 2008 Apr;79(4):433-9. doi: 10.3357/asem.2272.2008. PMID 18457303
- [Background] Ahmedzai S, Balfour-Lynn IM, Bewick T, Buchdahl R, Coker RK, Cummin AR, Gradwell DP, Howard L, Innes JA, Johnson AO, Lim E, Lim WS, McKinlay KP, Partridge MR, Popplestone M, Pozniak A, Robson A, Shovlin CL, Shrikrishna D, Simonds A, Tait P, Thomas M; British Thoracic Society Standards of Care Committee. Managing passengers with stable respiratory disease planning air travel: British Thoracic Society recommendations. Thorax. 2011 Sep;66 Suppl 1:i1-30. doi: 10.1136/thoraxjnl-2011-200295. No abstract available. PMID 21856702
- [Background] Lien D, Turner M. Recommendations for patients with chronic respiratory disease considering air travel: a statement from the Canadian Thoracic Society. Can Respir J. 1998 Mar-Apr;5(2):95-100. doi: 10.1155/1998/576501. PMID 9707451
- [Background] Aerospace Medical Association Medical Guidelines Task Force. Medical Guidelines for Airline Travel, 2nd ed. Aviat Space Environ Med. 2003 May;74(5 Suppl):A1-19. No abstract available. PMID 12817610
- [Background] Bradi AC, Faughnan ME, Stanbrook MB, Deschenes-Leek E, Chapman KR. Predicting the need for supplemental oxygen during airline flight in patients with chronic pulmonary disease: a comparison of predictive equations and altitude simulation. Can Respir J. 2009 Jul-Aug;16(4):119-24. doi: 10.1155/2009/371901. PMID 19707606
- [Background] Peckham D, Watson A, Pollard K, Etherington C, Conway SP. Predictors of desaturation during formal hypoxic challenge in adult patients with cystic fibrosis. J Cyst Fibros. 2002 Dec;1(4):281-6. doi: 10.1016/s1569-1993(02)00100-5. PMID 15463828
- [Background] Edvardsen A, Akero A, Christensen CC, Ryg M, Skjonsberg OH. Air travel and chronic obstructive pulmonary disease: a new algorithm for pre-flight evaluation. Thorax. 2012 Nov;67(11):964-9. doi: 10.1136/thoraxjnl-2012-201855. Epub 2012 Jul 5. PMID 22767877
- [Background] Edvardsen E, Akero A, Skjonsberg OH, Skrede B. Pre-flight evaluation of adult patients with cystic fibrosis: a cross-sectional study. BMC Res Notes. 2017 Feb 6;10(1):84. doi: 10.1186/s13104-017-2386-2. PMID 28166839